CLINICAL TRIAL: NCT05830916
Title: Diagnostic Role of Antiphospholipid Antibodies and Microparticles in Immune Thrombocytopenic Patients With Thrombosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SONagi, doctor, Assiut University
Other Study IDs: Thrombosis in ITP
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ITP with thrombosis: History taking including any medical history, family history, drug intake, arterial or venous thrombotic events.
  Venous blood samples will be collected by vein puncture under aseptic precautions for:
  Routine laboratory investigations:
  Complete blood picture with assessment of platelet count. Coagulation tests including prothrombin time (PT), activated partial thromboplastin time (APTT), fibrinogen and D-dimer.
  Liver and Kidney functions test.
  Specific laboratory investigations:
  Antiphospholipid antibodies assay which includes:
  Lupus anticoagulant (LA) by diluted Russel viper venom method. Anti β2glycoprotien І (β2GPІ), by enzyme-linked immunosorbent assay (ELISA). Anticardiolipin by (ELISA).
  Detection of Microparticles and their subtypes by flow cytometry:
  Annexin-v for all microparticles. CD 41 for platelet microparticles. CD 146 for endothelial microparticles.
  Interventions: Diagnostic Test: Antiphospholipid antibodies
- ITP without thrombosis: History taking including any medical history, family history, drug intake, arterial or venous thrombotic events.
  Venous blood samples will be collected by vein puncture under aseptic precautions for:
  Routine laboratory investigations:
  Complete blood picture with assessment of platelet count. Coagulation tests including prothrombin time (PT), activated partial thromboplastin time (APTT), fibrinogen and D-dimer.
  Liver and Kidney functions test.
  B- Specific laboratory investigations:
  Antiphospholipid antibodies assay which includes:
  Lupus anticoagulant (LA) by diluted Russel viper venom method. Anti β2glycoprotien І (β2GPІ), by enzyme-linked immunosorbent assay (ELISA). Anticardiolipin by (ELISA).
  Detection of Microparticles and their subtypes by flow cytometry:
  Annexin-v for all microparticles. CD 41 for platelet microparticles. CD 146 for endothelial microparticles.
  Interventions: Diagnostic Test: Antiphospholipid antibodies

INTERVENTIONS:
Diagnostic Test: Antiphospholipid antibodies — Antiphospholipid (aPL) antibodies are a heterogeneous group of autoantibodies with high affinity for phospholipids such lupus anticoagulant (LA), β2glycoprotien І (β2GPІ), and anticardiolipin (anti-CL). They interfere with physiological mechanisms of coagulation and fibrinolysis, leading the haemostatic balance towards coagulation. Moreover, it seems to affect the physiological function of various cells such as platelets and endothelial cells

SUMMARY:
Identify the procoagulant profile in immune thrombocytopenic patients with thrombosis.

Clinical implications of antiphospholipid antibodies in ITP patients with thrombosis.

Diagnostic role of microparticles in ITP patients with thrombosis.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an acquired autoimmune disorder characterized by isolated thrombocytopenia and an increased risk of bleeding. Paradoxically, ITP is also associated with an increased risk of thrombosis (1).

Recent studies showed that the occurrence of thrombosis in patients with ITP is not purely accidental and can be considered a clinical reality with an important impact on the management of the disease (2).

The pathophysiological mechanism for thrombosis in ITP remains unclear. Sever bleeding episodes are relatively rare in some patients with ITP although having low platelet count, suggests that these patients may have a protective factor against bleeding (3).

Antiphospholipid (aPL) antibodies are a heterogeneous group of autoantibodies with high affinity for phospholipids such lupus anticoagulant (LA), β2glycoprotien І (β2GPІ), and anticardiolipin (anti-CL). They interfere with physiological mechanisms of coagulation and fibrinolysis, leading the haemostatic balance towards coagulation. Moreover, it seems to affect the physiological function of various cells such as platelets and endothelial cells (4).

Microparticles (MPs) are a diverse group of bioactive small-sized vesicles (100-1000nm) that can be found in body fluids and blood after activation, necrosis, or apoptosis of almost all cells. Although most MPs in human blood originate from platelets, MPs are also released from leukocytes, erythrocytes, endothelial cells, smooth muscle cells and cancer cells (5). They participate in intercellular communication and play a major role in homeostasis under physiological conditions and also in diseases (6). The most prominent property of MPs is their procoagulant potential, mainly based on phosphatidylserine exposure and tissue factor expression (7).

Elevated levels of antiphospholipid antibodies and microparticles have been reported as a risk for development of prothrombotic state (8).

ELIGIBILITY:
Patients with confirmed diagnosis of primary chronic ITP with and without thrombosis, male or female above age of 18.Inclusion Criteria:

Exclusion Criteria:

Thrombocytopenic patients due to secondary causes such as pregnant women, patients with uncontrolled hypertension, peripheral or coronary artery disease, abnormal hepatic or renal function tests, bleeding disorder, and thrombopathy well be excluded from the study.

Patients full fill the criteria of antiphospholipid syndrome (APS).

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include 35 cases of ITP without thrombosis and 35 case of ITP with thrombosis.
  The sample size was calculated based on determining the main outcome variable using G*power software 3.1.9.2. based on the following assumption:
  Main outcome variable is difference between procoagulant profile of ITP patients with and without thrombosis especially for levels of antiphospholipid antibodies and microparticles (9).
  Main statistical test is one-sided student t-test to detect the difference between groups.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Identify the procoagulant profile in immune thrombocytopenic patients with thrombosis. | 2 years
  Clinical implications of antiphospholipid antibodies in ITP patients with thrombosis.
  Diagnostic role of microparticles in ITP patients with thrombosis.

REFERENCES:
- [Background] Rodeghiero F. ITP and thrombosis: an intriguing association. Blood Adv. 2017 Nov 14;1(24):2280. doi: 10.1182/bloodadvances.2017007989. eCollection 2017 Nov 14. No abstract available. PMID 29296876
- [Background] Boulware R, Refaai MA. Why do patients with immune thrombocytopenia (ITP) experience lower bleeding events despite thrombocytopenia? Thromb Res. 2020 Mar;187:154-158. doi: 10.1016/j.thromres.2020.01.020. Epub 2020 Jan 15. PMID 32004875
- [Background] Tomasello R, Giordano G, Romano F, Vaccarino F, Siragusa S, Lucchesi A, Napolitano M. Immune Thrombocytopenia in Antiphospholipid Syndrome: Is It Primary or Secondary? Biomedicines. 2021 Sep 6;9(9):1170. doi: 10.3390/biomedicines9091170. PMID 34572358
- [Background] Reid VL, Webster NR. Role of microparticles in sepsis. Br J Anaesth. 2012 Oct;109(4):503-13. doi: 10.1093/bja/aes321. Epub 2012 Sep 4. PMID 22952169
- [Background] Nomura S, Shimizu M. Clinical significance of procoagulant microparticles. J Intensive Care. 2015 Jan 7;3(1):2. doi: 10.1186/s40560-014-0066-z. eCollection 2015. PMID 25705427
- [Background] Chaturvedi S, Cockrell E, Espinola R, Hsi L, Fulton S, Khan M, Li L, Fonseca F, Kundu S, McCrae KR. Circulating microparticles in patients with antiphospholipid antibodies: characterization and associations. Thromb Res. 2015 Jan;135(1):102-8. doi: 10.1016/j.thromres.2014.11.011. Epub 2014 Nov 15. PMID 25467081
- [Background] Alvarez-Roman MT, Fernandez-Bello I, Jimenez-Yuste V, Martin-Salces M, Arias-Salgado EG, Rivas Pollmar MI, Justo Sanz R, Butta NV. Procoagulant profile in patients with immune thrombocytopenia. Br J Haematol. 2016 Dec;175(5):925-934. doi: 10.1111/bjh.14412. Epub 2016 Oct 21. PMID 27766635